CLINICAL TRIAL: NCT06747442
Title: Culturally Engaged REcovery - MOms Connected Through Native CommunitY (CEREMONY)
Brief Title: Culturally Engaged REcovery: MOms Connected Through Native CommunitY
Acronym: CEREMONY
Status: Not yet recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michelle Debbink, Assistant Professor, University of Utah
Other Study IDs: 00177269; U54HD113169 (NIH)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Substance Use Disorders (SUD); Pregnancy; Maternal Morbidity and Mortality; Cultural Adaptation
Keywords: Pregnancy; Prenatal care; Substance Use Disorder; Native and Indigenous Health; Culturally adapted care
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CEREMONY: Any Native individuals seeking treatment in the integrated perinatal SUD clinical program specifically created for Native mothers may opt to enroll in prospective data collection during their time in the program
- Contemporary comparison cohort: Utah Population Database will be queried for individuals who could have met criteria for prospective data collection but did not participate in the SUD clinical program. The outcomes of these individuals (administrative data only) will be compared to individuals taking part in the SUD program for Native pregnant people who agree to have their data collected.

SUMMARY:
Pregnant and postpartum American Indian and Alaska Native people (Native mothers) face a more than two-fold higher risk of maternal mortality compared to non-Hispanic White mothers. Deaths related to substance use (SU) and mental health conditions are a leading cause of preventable maternal mortality, including among Native mothers, making these conditions a strong target for reducing maternal mortality and morbidity. The objective of our study is to 1) adapt evidence-based perinatal care models that integrate pregnancy and postpartum care with SU treatment and care to meet the needs of Native mothers, and 2) assess the implementation and efficacy of that model for participants with substance use disorder who identify as Native receiving prenatal care at Sacred Circle Healthcare in Salt Lake City, Utah.

DETAILED DESCRIPTION:
Pregnant and postpartum American Indian and Alaska Native people (Native mothers) face a more than two-fold higher risk of maternal mortality compared to non-Hispanic White mothers. Deaths related to substance use (SU) and mental health conditions reflect a leading cause of preventable maternal mortality, including among Native mothers, making these conditions a strong target for reducing maternal mortality and morbidity. The Utah Maternal Mortality Review Committee (MMRC) has identified access to substance use disorder (SUD) treatment including medication for opioid use disorder (MOUD), mental health care, improved social support, decreased stigma against SUD, and care coordination, particularly in the postpartum period (when the majority of deaths occur) as actionable intervention points. The objective of our study, Culturally-Engaged REcovery - MOms connected through Native CommunitY (CEREMONY), is to adapt evidence-based perinatal care models that integrate pregnancy and postpartum care with SU/SUD treatment and care to meet the needs of Native mothers. With our partners at Sacred Circle Clinic, a federal Tribal Contract clinic operated by the Confederated Tribes of the Goshute Reservation, we are uniquely poised to respond to the expressed needs of Native mothers and stakeholders, who identified a lack of culturally-integrated SUD care as a significant gap in perinatal care for Native mothers. We will do this by building upon the strong, evidence-based foundation of our University of Utah integrated perinatal SUD clinic called Substance Use and Pregnancy - Recovery, Addiction, and Dependence (SUPeRAD). The SUPeRAD model directly addresses the actionable intervention points identified by the MMRC to prevent SUD-related maternal deaths, but is not specifically adapted to Native mothers' needs. The rationale for this study is that there is a critical knowledge gap in the adaptation and implementation of integrated perinatal SUD care specifically for Native mothers. The CEREMONY study will fill this gap by adapting the SUPeRAD clinic model to the needs of Native mothers using the validated ADAPT-ITT adaptation framework, informed by human centered design and community-based participatory research (Aim 1; not part of the observation trial submission described on this website); and then studying the adapted, culturally-integrated perinatal SUD care intervention at Sacred Circle Healthcare using a Hybrid Type 1 effectiveness-implementation study (Aim 2a&b). The Hybrid Type 1 design will provide important, reliable data on the clinical effectiveness of culturally adapted perinatal SUD care for Native mothers (Aim 2a) while also producing novel data on the implementation process (Aim 2b). Successful completion of these Aims will provide implementation and training protocols that can be used to guide adaptation and implementation of culturally-adapted perinatal SUD care in other settings across the US.

Sacred Circle Healthcare will be implementing the new care model and offering it to all patients who identify as Native and having a substance use disorder. Within that group, the CEREMONY study will invite patients who meet study inclusion criteria to participate in the observational research study.

Participants enrolled prospectively will be compared to a historical cohort, with data pulled from the Utah Population Database, for our primary outcome. The historical cohort will be comprised on deidentified data from individuals over 18 years old with delivery of an infant greater than 20 weeks' gestation between 2020 and the most recent year of available data (approximately 2027-28) who had at least one visit with a Utah health provider before delivery and identify as American Indian/Alaska Native based on vital records or hospital records.

ELIGIBILITY:
CEREMONY Inclusion Criteria:

* English or Spanish speaking
* pregnant (verified by point of care urine pregnancy test)
* plan to carry the fetus to delivery
* identify as Indigenous, Native, Native American, American Indian or Alaska Native
* willing to grant a release of information to allow study staff to contact other health care institutions and treatment centers and collect information from the medical record, e.g., date of delivery, infant admission etc.

CEREMONY Exclusion Criteria:

* have a documented psychotic episode in the last 30 days
* be >39 weeks of gestation
* be unable provide collateral contact information of at least 1 person
* be unable to provide reliable phone number
* plan to move within 3 months of delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study compares the outcomes of two groups: 1) Native individuals who have decided to participate in a new clinical program for pregnant Native mothers with SUD (program cohort) who then also agree to have their data to collected prospectively; and 2) pregnant Native mothers with SUD identified through administrative data who did not participate in the clinical program. The study population as a whole consists of Native and Indigenous pregnant individuals with SUD in the state of Utah.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Postpartum engagement in care | From enrollment until 12 weeks after delivery
  Completion of a postpartum follow up visit within 8 weeks of delivery

SECONDARY OUTCOMES:
Medication for opioid use disorder | Enrollment through 1 year postpartum
  Any prescription of suboxone or methadone for individuals with OUD, and the length of time the prescription is kept current

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Debbink, MD PhD, Principal Investigator — University of Utah; Adam Gordon, MD, Principal Investigator — University of Utah
Locations (1):
- Sacred Circle Healthcare, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Data sovereignty is of critical importance when working with Native communities. Particularly with recent data breaches in Utah related to Native individuals' health data, a clear and strictly adhered-to data management policy is critical. The memorandum of understanding between the University of Utah and Sacred Circle includes a data sovereignty plan, which includes a statement that data is owned by the Tribal entity. Data will be deidentified before sharing on a need to know basis, on the agreement that once the data analysis is complete, the data will be returned to the Tribal entity or destroyed.

REFERENCES:
- [Derived] Debbink MP, Tanana H, Murray JL, Blosser P, Horse L, Monroy C, Spiess S, Charles JE, Turok DK, Smid MC, Allshouse AA, Smith JD, Cohen SR, Johnson EP, Metz TD, Gordon AJ. Culturally Engaged REcovery - MOms connected through Native CommunitY (CEREMONY): An Implementation Study to Evaluate the Adaptation and Implementation of an Integrated Perinatal SUD Clinical Model for Pregnant and Postpartum Native People. Subst Use Addctn J. 2026 Jan;47(1):233-242. doi: 10.1177/29767342251336550. Epub 2025 Sep 15. PMID 40955087